CLINICAL TRIAL: NCT03651843
Title: Perception of Risks Into Work During Pregnancy Among Post-partum Women in the Lille Metropolis
Acronym: PERISTRAG
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017_88; 2018-A00962-53 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-08-01; First posted 2018-08-29 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Pregnancy, High Risk
Keywords: high risk; pregnant women; occupational hazard; occupational risk
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy subjects
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Women who have recently given birth in the Lille metropolitan area fill in a self-administered questionnaire asking them about their perception of occupational risk during pregnancy and their knowledge of their right to work during pregnancy.
  Other Names: Occupational risk exposure questionnaire during pregnancy

SUMMARY:
In ten years, the labor force has grown by 1.4 million people according to French national institute for statistical and economic studies. This increase is partly due to the increased presence of women in the labor market. Thus, the majority of some 800,000 annual births come from working women. However, some women in professional activity may be exposed to occupational risks, which may have effects on the develop-ment of the fetus during pregnancy. France benefits from protective legislative measures against pregnant women. Recommendations already exist.

But with medical desertification, pregnant women may have more difficulty contacting their occupational doctor or treating physician and to access information about the risks to her work-related pregnancy.

It seems to us important to be able to better quantify the information needs of women in this problem.

ELIGIBILITY:
Inclusion Criteria:

* working during their pregnancy (at least 2 months, including the beginning of pregnancy
* having given birth during the period of inclusion
* in a hospital or clinic of Lille metropolis volunteer to participate in the study

Exclusion Criteria:

* minor women
* unemployed
* student
* guardianship
* work abroad
* change of employer during pregnancy
* inability to answer the questionnaire

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women who have just given birth in maternity hospitals in the Lille metropolis and who worked during their pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
percentage of women who thought they had occupational exposures at risk for their baby during pregnancy | At childbirth
  the different occupational exposures are listed. If the woman has been exposed and thinks it's dangerous for her baby, she reports it.

SECONDARY OUTCOMES:
adaptation or not of the workstation in case of exposure to a professional risk | at childbirth
  if the woman is exposed to a defined risk and her job has been set up to avoid this risk during pregnancy, she reports it
percentage of women with a score of at least 5 out of 10 | at childbirth
  knowledge of French legislation concerning the protection of pregnant women at work of current legislation referenced in a questionnaire that includes 10 binary questions. A score will be calculated by summing the answers (score out of 10)

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Fantoni, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Claude Huriez, CHU, Lille, France